CLINICAL TRIAL: NCT06396624
Title: Effects of Photobiomodulation on the Innate Immune System of Neonates and Infants Diagnosed With Acute Respiratory Sintitial Virus Bronchiolitis - Randomized Controlled Trial
Brief Title: Effects of Photobiomodulation on the Innate Immune System of Neonates and Infants With Bronchiolitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MazzoDM_PHD_FurlanettoKC
Record Dates: First submitted 2024-01-18; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Bronchiolitis; Virus; Virus Disease
Keywords: Bronchiolitis; Photobiomodulation; Low Level Light Therapy; Children
MeSH Terms: conditions — Bronchiolitis; Virus Diseases | interventions — Low-Level Light Therapy; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The application of FBM will take place immediately after the conventional physical therapy maneuvers as recommended by the institution's physical therapist, following the institution's protocols. The patient may be positioned in bed or on the lap of the person in charge, in the way that is most comfortable for him/her, with the chest bare. The eyes of the patient, the person in charge and the physiotherapist must be properly protected by the use of appropriate glasses to avoid contact with the light beam emitted by the equipment. The application will be punctual, perpendicular to the thorax, using the portable photobiomodulation device Therapy EC - (DMC equipamentos - São Carlos-SP. ANVISA Registration: 80030819013) in continuous mode, with a power of 100mW, 808nm wavelenght, 4J of energy and 40s of irradiation per point.
  Interventions: Radiation: Intervention Group photobiomodulation
- Control Group (Placebo Comparator): The control group will be treated in the same way as the intervention group, as recommended by the institution's physiotherapist, following its protocols. The same photobiomodulation device will be used as a placebo, but turned off, with a lock on the tip to ensure that no light beam is emitted. The device will be wrapped in PVC plastic film that allows it to be cleaned and changed when used in different patients, avoiding possible contamination. The same irradiation points will be used as in the control group (Figures 2 and 3). The patient may be positioned in bed or on the lap of the person in charge, in the way that is most comfortable for him/her, with the chest bare. The eyes of the patient, the caregiver and the physiotherapist must be properly protected.
  Interventions: Other: Control Group

INTERVENTIONS:
Radiation: Intervention Group photobiomodulation — Seven spots on child's thorax and two spots on the face will be irradiated with 40s per point of photobiomodulation.
  Other Names: Photobiomodulation; Low level light therapy; Low level laser
  Arms: Intervention Group
Other: Control Group — The photobiomodulation device will positioned in seven spots on thorax and two in child's face, but it will not emit any time of radiation, since the device will be turned off.
  Arms: Control Group

SUMMARY:
The innate immune response of children with acute viral bronchiolitis (AVB) caused by respiratory syncytial virus (RSV) in the acute phase and in the resolution phase, is marked by variations in inflammatory and anti-inflammatory mediators, where in the acute phase there is recruitment and activation of multiple cells of the immune system, with consequent increase in the expression of pro-inflammatory mediators. Evidence indicates that there is a considerable increase in tumor necrosis factor-alpha (TNF) , interleukine 6 (IL6), interleukine 1-beta, interleukine 8 (IL8) interleukine 10 (IL10), exposing to IL6, IL8 and IL-10 positively correlated with AVB severity. There are already reports that the transcutaneous application of photobiomodulation (PBM) reaches the lungs, producing positive responses in respiratory pathologies, both acute and chronic . Thus, PBM caused by the use of low-level laser may be a favorable resource to be used in the area of respiratory physiotherapy, specifically in neonatology and pediatrics, since there are studies in both experimental and human models that prove its action on lung cells, acting to reduce airway edema, reduce neutrophil migration to lung tissue and synthesize pro-inflammatory cytokines TNFalpha, IL6 and IL-10. In addition, it is a portable, practical, quick application, with minimal contraindications and possibly better tolerated by the neonatal and pediatric population.

DETAILED DESCRIPTION:
Acute Viral Bronchiolitis (AVB) is the most common disease of the lower respiratory tract in children, being one of the major causes of hospitalization in children under two years of age, especially in winter. It is characterized by inflammation, edema, and necrosis of cells of the small airways epithelium, with increased mucus secretion and bronchospasm. Among the most common pathogens for the development of AVB are rhinovirus, influenza A and B, parainfluenza, metapneumovirus, adenovirus, however, the most common and responsible for 70% of AVB in children under two years of age is respiratory syncytial virus (RSV). RSV is highly contagious and infectious, accounting for 2-3% of the hospitalization of infected children, and there is a seasonal variation in RSV infection levels, which are higher during the winter in temperate regions, and this occurs because low temperatures and high humidity favor the proliferation of the virus.

RSV is transmitted through the air in contact with the nasal epithelium, mouth, eyes, or contaminated surfaces, and the incubation time is three to eight days. As soon as the virus reaches the nose or mouth, it begins to infect the epithelial cells of the upper respiratory tract, then progresses to the lower airways reaching the bronchioles where it replicates more easily, thus developing bronchiolitis. Inflammation and obstruction of the bronchioles then occurs, resulting in reduced airflow in the small caliber airways, altering the ability to exhale, which leads to hyperinflation, increased mucus production, atelectasis and wheezing. Immunopathology occurs through the expression of pro-inflammatory cytokines with subsequent perivascular and peribronchial infiltration of mononuclear cells, mostly neutrophils and lymphocytes, triggering an unbalanced response between T helper cells 1 and 2.

In addition to AVB, RSV infection can lead to pneumonia in addition to the possibility of later development of wheezing and asthma, so there is growing concern about how RSV infections in the first months of life can lead to the development of chronic lung diseases. in addition to being considered the second pathogenic agent causing death in children under one year of age.

The inability of the innate immune system of neonates and children to fight RSV infection and its serious consequences makes the development of new prevention and treatment strategies a priority.

To meet this need, notable advances have been made in recent years in relation to low-level laser PBM applied to lung diseases. PBM is a non-invasive, adverse-effect-free, accessible, and well-tolerated resource for patients diagnosed with pulmonary diseases such as chronic obstructive pulmonary disease, COVID-19 and asthma. Many effects are attributed to PBM and one of the main ones is its antioxidant and anti-inflammatory effects at the cellular level. From the penetration of the photon into the tissue where it interacts with intracellular molecules and initiates a series of changes in its functioning, including membrane permeability and cellular metabolism, regulating antioxidative defenses and reducing oxidative stress.

Jahani-Sherafat et al. (2020) in their review explain the various hypotheses for PBM in cellular functions, the first refers to cytochrome-c oxidase, obtained by infrared light. Other hypotheses are that photons separate nitric oxide from the enzyme and make this nitric oxide active and increase electron transport, mitochondrial membrane potential, and adenosine triphosphate (ATP) production. Another hypothesis is related to light-sensitive ion channels that can lead to the accumulation of calcium in cells, and after photon absorption, several signaling channels are activated using reactive oxygen species, cyclic adenosine monophosphate (AMP), nitric oxide, and calcium, leading to the stimulation of transcription factors. With these factors activated, the expression gene increases and as a result, increases protein synthesis and proliferation, anti-inflammatory signaling, anti-apoptotic proteins, and antioxidant enzymes.

Scientific studies, both in animal and human models, has been developed focused on reducing inflammatory conditions resulting from both acute and chronic respiratory pathologies. In general, these studies demonstrate that the transcutaneous application of PBM reaches the lungs and positively interferes with inflammatory and immunological processes in lung lesions. It can be a viable resource as an adjuvant in the treatment of respiratory pathologies.

Study Design:

The study will be a randomized clinical trial and the sample consisted of neonates and infants from zero to 24 months of age, diagnosed with AVB hospitalized at the Maternal and Child University Hospital of the Universidade Estadual de Ponta Grossa. The project will be submitted for approval by the Human Research Ethics Committee, and subsequently registered in the ClinicalTrials.gov database.

The parents or guardians of the newborn or infant will be invited to participate in the study and, if they are interested, they must consent to participate by signing the free and informed consent form. The purpose of the study will be explained to those responsible and they will be able to ask questions at any time about the procedures to be performed. If the parents or guardians wish to leave the study, there will be no harm to the patient's treatment, which will be as established in the randomization.

The admission of patients diagnosed with AVB to the participating hospitals will be checked daily. As soon as the patient is identified, in the first physical therapy consultation, the person in charge will be invited to participate in the research through the informed consent form. If accepted, the physiotherapist will proceed with the questions on the follow-up form, after which the physiotherapy will follow the physiotherapy service according to the indicated randomization. In this first consultation, the International Study of Wheezing (EISL) questionnaire will be applied, AVB severity will be determined by the Wang scale, and tracheal secretion samples will be collected. The results of routine laboratory tests will be monitored daily to record the values. A new sample of tracheal secretion will be collected on the fourth day of hospitalization, the last sample will be collected on the eighth day of hospitalization or earlier if the patient is discharged from the hospital. For follow-up, the researcher will contact the parents or guardians after completing three months of hospital discharge to apply a questionnaire prepared by the author that will contain the following questions: How many times has your child had a cold/flu in the last few months?; If so, did he/she needed to be hospitalized?; Are your child's vaccinations up to date?; Did your child start attending daycare or school during this period?; Has there been a change in the child's diet? (e.g. food transition); Do you notice your child tired to play?

Randomization and blinding:

Randomization will be done in blocks and generated by a computer program, being concealed in sealed and sequentially numbered opaque envelopes, implemented by someone who has no involvement in the study. Each envelope will correspond to one of the two study groups and an envelope will be chosen by the participant's guardian at the time of evaluation. The statistical evaluator will be blinded to the allocation of patients into the groups.

* Sample Calculation In order to reject the null hypothesis, it is estimated that 18 participants will be needed in each group with a sample power of 95% and a value of p<0.05, however, estimating a possible loss of 20% over the course of the study, the sample size will be 22 individuals in each group. The calculation was based on the study by Mehani (2017), who analyzed the values of interleukin IL6 in a group of adults with chronic obstructive pulmonary disease who were treated with FBM compared to a group treated with respiratory exercisers, where the final mean IL6 in the PBM group was 49.4(10.1) and in the exerciser group it was 62.8(11.4) with a value of P<0.0001.
* Statistical analysis Data tabulation will be performed using Microsoft Excel and statistical analysis using SPSS 22.0 and GraphPad Prism 6.0. The verification of the normality of the data will be performed by the Kolmogorov-Smirnov test. Variables with normal distribution will be presented as mean ± standard deviation, variables with non-normal distribution will be presented as median and interquartile range 25-75%, and categorical variables will be presented as absolute and relative frequency. To identify the effects of FBM on BVA, the mixed repeated measures ANOVA test will be used. The intra-group factor will be the allocation group (control group or intervention group) and the intra-group factor will be the moment of evaluation (D1 and Dalta for laboratory tests and Wang score; D1, D4 and D8/or discharge for tracheal discharge). Statistical significance will be determined as P<0.05. The follow-up questionnaires will be compared using the non-parametric Student's t-test or the Mann-Whitney test according to the normality of the data.

Due to its originality, this study has great potential for publication in renowned scientific journals. If the hypothesis that MBF promotes the reduction of cellular inflammatory status is confirmed, the benefits will be related to a shorter hospital stay, faster resolution of the lung infection, in addition to consolidating MBF as another effective resource in the respiratory physiotherapy action in the treatment of AVB in this population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AVB due to RSV confirmed on hospital admission examination

Exclusion Criteria:

* Diagnosis of congenital or acquired heart disease;

  * Pulmonary malformations;
  * Use of any number of doses of palivizumab or another immunobiological agent;
  * Present any "new pathology" during treatment with FBM;
  * Cancer of any histology;
  * Skin lesion near the application sites;
  * Desire to drop out of study.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-06-18 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Innate Immunological Markers | 4th day of hospitalization and 8th or discharge day
  Due to the increase in nasotracheal secretion caused by AVB, nasotracheal aspiration is usually a routine procedure because it is often necessary to perform it to maintain the pervious airways, since in some cases children cannot properly manage the secretion. Thus, this procedure will be used to collect secretion on the first, fourth and eighth days of care, stored in a -80°C freezer and later sent for laboratory analysis of pro-inflammatory cytokines such as: tumor necrosis factor alpha (TNF), interleukin 6 (IL6), interleukin 1-beta, and anti-inflammatory interleukin 10 (IL10). Cytokine analysis will be performed by flow cytometry using the BD™ Cytometric Bead Array (CBA) kit.

SECONDARY OUTCOMES:
Severity of AVB | 1st day of hospitalization through 8th or discharge day
  To assess the severity of AVB, the Wang score will be used, which evaluates four items: respiratory rate, presence of wheezing, presence of chest retractions, and general condition. The sum of the items generates a value from zero to 12, classifying AVB as mild, moderate and severe, with 12 being the greatest severity of the disease (WANG et al. 1992). This scale will be applied daily before physical therapy care during the hospitalization period in all participants. Along with the scale, the following will be recorded: respiratory rate, heart rate, temperature, peripheral O2 saturation, type oxygen therapy (interface and flow).
Overall | 1st day of hospitalization through 8th or discharge day
  General data will be collected, in a Google form (Google Corp. 2018), such as: current age, gestational age at birth, type of delivery, gender, duration of exclusive breastfeeding, previous diagnosis of respiratory diseases, previous hospitalizations, time and place of hospitalization (emergency room, ward, intensive care unit), use and time of use of oxygen therapy, use and time of use of invasive and/or non-invasive mechanical ventilation, if attending a daycare center or school, concomitant infection by other respiratory viruses, clinical picture, onset of symptoms, date of hospitalization and start of FBM application, skin color (phototype), presence of jaundice, total number of FBM applications, total number of physical therapy visits, medications used during hospitalization and medications used continuously at home.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Pesquisa e Pós Graduação na Unopar, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No